CLINICAL TRIAL: NCT06100263
Title: Breast Cancer Resiliency Through Exercise Program (B-REP): Pilot Study
Brief Title: Breast Cancer Resiliency Through Exercise Program (B-REP)
Acronym: B-REP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UMCC 2023.092; HUM00244376 (Other: University of Michigan)
Record Dates: First submitted 2023-10-20; First posted 2023-10-25 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Supervised exercise) (Experimental): The individualized program is based on participants' baseline 5-repetition maximum muscular strength assessment and is aligned with current cancer-specific exercise recommendations. The resistance program will follow the FITT principle (frequency, intensity, time, and type):
  Frequency. Participants will aim for 3 resistance exercise sessions per week. Intensity. Resistance exercise intensity will have a schedule for increased progression by both load via increased weight and volume via increased repetitions and sets. If participants are not able to increase resistance loads as scheduled, they will remain at their current load and volume until the next scheduled increase.
  50% of 5-repetition maximum for upper and lower body. 3 sets of 8 to 12 repetitions.
  60% of 5-repetition maximum for upper and lower body. 3 sets of 8 to 12 repetitions.
  70% of 5-repetition maximum for upper and lower body. 4 sets of 8 to 12 repetitions.
  Interventions: Other: Individualized exercise program
- Control (waitlist) (Active Comparator): Participants randomized to the waitlist control condition will be on a waiting list for 24 weeks. Participants in waitlist control condition will complete measures on the same schedule as intervention participants. After 24 weeks, participants will be offered to participate in the online sessions with an exercise trainer using Zoom twice per week for 12- weeks. The sessions will be 30 to 45minutes in length.
  Interventions: Other: Control Arm

INTERVENTIONS:
Other: Individualized exercise program — guided exercise program for 12 weeks
  Arms: Intervention (Supervised exercise)
Other: Control Arm — Control Arm Waiting List for 24 weeks, then offered a guided exercise program for 12 weeks
  Arms: Control (waitlist)

SUMMARY:
The study will use a cross-sectional study design with a follow-up 2-arm randomized controlled trial with that has assessments at baseline, post-intervention (i.e., Week 12), and 3-months post-intervention (i.e., Week 24). The 2 arms are the 12-week intervention and waitlist control among 30 Black breast cancer survivors

DETAILED DESCRIPTION:
14AUG2025- The sample size was updated, and the questionnaire was split into 2 questionnaires, as a planned solution in response to a low accrual

28OCT2025- Amendment was processed to update design and intervention items. The exercise threshold was changed from a 1-repeition maximum (1RM) to a 5-repeptition maximum (5RM). Since the intervention includes functional exercises, so we elected to use a functional strength (5RM) outcome rather than a maximal strength outcome (1RM) to better align with the intervention. The control condition was changed to a waitlist design. A waitlist control is more engaging, and there is a higher likelihood of retaining control participants.

ELIGIBILITY:
Inclusion Criteria:

Women will be eligible if they meet the following criteria:

* self-identify as Black or African American or Afro-Latina/e;
* are ≥18 years old;
* have a confirmed diagnosis of breast cancer, Stage I to IIIA;
* have completed primary active treatment (i.e., surgery, chemotherapy, and radiation) within 5 years prior to study start where concomitant hormonal therapy is acceptable;
* are not meeting current cancer-specific resistance exercise guidelines of ≥ 2 times per week; and
* are able to speak and understand English.

Exclusion Criteria:

* metastatic disease;
* medical reason that precludes them from increasing current exercise levels;
* planned elective surgery during study period;
* pregnant or plans to become pregnant during the study period;
* plans to move out of United States during the study period; (the rationale for this exclusion is that it will be difficult to conduct the in-person assessments if a participant leaves the United States);
* current enrollment in another exercise trial; and/or
* inability to pass exercise pre-screening or receive physician consent to increase current physical activity levels.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the exercise program (Retention) | up to 24 weeks after start of intervention
  Percent of patients that complete the intervention
Feasibility of the exercise program (Adherence) | 12 weeks after start of intervention
  Percent of patients that complete the exercise sessions
Feasibility of the exercise program (fidelity) | 12 weeks after start of intervention
  Upon completion of the trial, a random sample of 10 recorded sessions will be analyzed for fidelity. Research staff who did not conduct the intervention will use a "fidelity checklist" of specific exercises and intervention characteristics (e.g., allowing time for questions, cueing for proper posture and form, etc.) required for each exercise session..
Satisfaction of program | up to 24 weeks after start of intervention
  14-item scale measuring ease of use, convenience, engagement, enjoyment, and privacy elements of the intervention.
Affective attitude | up to 24 weeks after start of intervention
  36-item scale assessing views, attitude, and experiences in exercise87
Perceived burden | up to 24 weeks after start of intervention
  Single item, "Now that you've completed this part of the study, how burdensome or difficult did you find the experience. Select the response that best represents your experience." (1= Very burdensome to 5= Not too burdensome.)
Outcome expectation | up to 24 weeks after start of intervention
  15-item scale assessing physical, social, and self-evaluative outcomes of exercise

CONTACTS AND LOCATIONS:
Overall Officials: Angela Fong, PhD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No